CLINICAL TRIAL: NCT02597738
Title: Scientific and Methodological Advancements in Human Specimens to Further the Development of Lung Cancer-based Precision Medicine - A Feasibility Study
Brief Title: A Feasibility Study to Further the Development of Lung Cancer-based Precision Medicine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 204803
Record Dates: First submitted 2015-10-28; First posted 2015-11-05 (Estimated); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer; Head and Neck Cancer
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Lung/ Head and Neck Cancer Group (Experimental): Blood/Urine Sample Collection Fresh tissue biopsy A one time fresh tissue biopsy of the patient's lung cancer (outside of their normal standard of care biopsy) will be collected for the research. Patients will also complete research blood and urine sample collections every two to four weeks for one year, then up to 120 days for years two through five.
  Interventions: Other: Fresh tissue biopsy; Other: Blood/Urine Sample Collection
- Chronic inflammatory disease (Experimental): Blood/Urine Sample Collection A one time blood and urine sample collection will be completed.
  Interventions: Other: Blood/Urine Sample Collection
- At risk for lung cancer (Experimental): Blood/Urine Sample Collection A one time blood and urine sample collection will be completed.
  Interventions: Other: Blood/Urine Sample Collection
- Healthy people who exercise (Experimental): Blood/Urine Sample Collection Blood and urine collection one time prior to exercise and one time after exercise.
  Interventions: Other: Blood/Urine Sample Collection
- Lung cancer with planned resection (Experimental): Blood/Urine Sample Collection Blood and/or urine sample collection one time before surgery and one time after surgery. Blood and/or urine sample collection at subsequent visits.
  Fresh tissue biopsy Tissue sample collection from surgery is there is any tissue considered to be pathological waste that would normally be discarded.
  Interventions: Other: Fresh tissue biopsy; Other: Blood/Urine Sample Collection
- Solid tumor cancer w/ radiation therapy (Experimental): Blood/Urine Sample Collection Blood and/or urine sample collection prior to radiation treatment. Blood and/or urine collection after completion of radiation therapy. Blood and/or urine collection at subsequent visits for next 5 years.
  Interventions: Other: Blood/Urine Sample Collection

INTERVENTIONS:
Other: Fresh tissue biopsy — Fresh tissue biopsy will be collected.
  Arms: Lung cancer with planned resection; Lung/ Head and Neck Cancer Group
Other: Blood/Urine Sample Collection — A one time blood sample will be collected.

SUMMARY:
The purpose of this study is to further advancements in biospecimens (blood cellular free component, e.g., plasma, serum, tissue, urine), in order to develop precision medicine, for lung cancer management and lung cancer screening (synergy with imaging). A co-clinical trial approach, with integrative analyses leveraging data from the treatment of genetic mouse models of lung cancer along with clinical samples and data from lung cancer patients, will be used to elucidate genomic background metrics, identify cell free DNA mutations, and further refine the liquid biopsy approach. Blood and urine samples will be analyzed for different genetic components. The tissue biopsy will be implanted into a mouse and after the cancer grows in the mouse the cancer DNA from the mouse will be compared with the human blood.

DETAILED DESCRIPTION:
This is a feasibility study to collect tumor and peripheral blood and urine of patients with lung cancer, or head and neck cancer, or other solid tumor who receive treatment. Blood and urine will also be collected from subjects without cancer to assess non cancer profiles. To conduct this study, a total of 30 study-eligible subjects of all races and ethnicities, aged 18 years or older with a diagnosis of cancer of the lung or head and neck cancer or other solid tumor malignancy (Cohort A), will be enrolled and have their tumor collected once for molecular profiling and xenograft development and blood collected at prespecified time intervals until completion of treatment for liquid biopsy analysis (targeted sequencing, whole exome sequencing, whole genome sequencing). A total of 140 study-eligible subjects of all races and ethnicities ages 18 years or older will be enrolled in the non-lung cancer control subgroups for chronic inflammatory disorder (Cohort B), people at risk to develop lung cancer (Cohort C) and healthy people who complete vigorous exercise (Cohort D). A total of 180 subjects will be enrolled into the resection and radiation therapy cancer cohorts (Cohorts E and F).

ELIGIBILITY:
Cohort A (Lung/Head and Neck Cancer Group) Inclusion criteria:

1. Unresectable metastatic lung cancer or head and neck cancer or other solid tumor malignancy
2. Current or Former Smokers with greater than or equal to 10 pack year smoking history
3. Candidates for standard or experimental treatment as determined by their treating physician
4. Age 18 years and older
5. Must sign an informed consent approved by the UAMS Institutional Review Board (IRB)

Cohort A (Lung/Head and Neck Cancer Group) Exclusion criteria:

1. Any other significant medical or psychiatric conditions which, in the opinion of the enrolling investigator, may interfere with consent or compliance of the treatment regimen
2. Existing diagnosis or evidence of Hepatits C, Rheumatoid Arthritis or any previous solid organ transplant.
3. Existing diagnosis or evidence of organic brain syndrome that might preclude participation in the full protocol
4. Existing diagnosis or history of significant impairment of basal cognitive function that might preclude participation in the full protocol
5. Other significant medical or psychiatric conditions which, in the opinion of the enrolling investigator, may interfere with consent or compliance of the treatment regimen

Cohort B (Chronic Inflammatory disease) Inclusion criteria:

1. Chronic inflammatory disease including but not limited to:

   * Systematic Lupus Erythematosus
   * Rheumatoid arthritis
   * Hepatitis C
   * Ankylosing Sponsylitis
   * Scleroderma
2. No history of smoking or quit smoking within the last six months
3. Age 18 years and older
4. Must sign an informed consent approved by the UAMS Institutional Review Board (IRB)

Cohort B (Chronic inflammatory disease) Exclusion criteria:

1. Any other significant medical or psychiatric conditions which, in the opinion of the enrolling investigator, may interfere with consent or compliance of the treatment regimen. 2. Existing diagnosis or evidence of organic brain syndrome that might preclude participation in the full protocol.

3. Existing diagnosis or history of significant impairment of basal cognitive function that might preclude participation in the full protocol.

4. Other current malignancy(s). Subjects with prior history at any time of any in situ cancer, including lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ or basal or squamous skin cancer are eligible, provided they are disease-free at the time of registration. Subjects with other malignancies are eligible if they have been continuously disease free for ≥ 5 years prior to the time of registration.

5. No current steroid treatment or treatment within the last 3 months.

Cohort C (At risk for lung cancer) Inclusion criteria:

1. Age 45-74 years
2. Former or current smokers with a 30 or more pack-years of cigarette smoking history
3. Must sign an informed consent approved by the UAMS Institutional Review Board (IRB)

Cohort C (At risk for lung cancer) Exclusion criteria:

1. Other current malignancy(s). Subjects with prior history at any time of any in situ cancer, including lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ or basal or squamous skin cancer are eligible, provided they are disease-free at the time of registration. Subjects with other malignancies are eligible if they have been continuously disease free for ≥ 5 years prior to the time of registration.
2. History of lung cancer
3. History of removal of any portion of the lung, excluding needle biopsy
4. Unexplained weight loss of more than 15 pounds in the 12 months prior to eligibility assessment
5. Recent hemoptysis
6. Pneumonia or acute respiratory infection treated with antibiotics in the 12 weeks prior to eligibility assessment.
7. History of abnormal chest CT examination suspicious for cancer in the 18 months prior to eligibility assessment.

9. Chronic inflammatory disease including but not limited to:

* Systematic Lupus Erythematosus
* Rheumatoid arthritis
* Hepatitis C
* Ankylosing Sponsylitis
* Scleroderma

Cohort D (healthy people who exercise) Inclusion criteria:

1. Age 18 years and older
2. Must sign an informed consent approved by the UAMS Institutional Review Board (IRB)
3. Must complete and self-report vigorous exercise for 30 minutes

Cohort D (healthy people who exercise) Exclusion criteria:

1. People will be excluded if they have self reported any of the following conditions: diabetes, heart disease, autoimmune disorders or hepatitis.

Cohort E (lung cancer with planned resection) Inclusion criteria:

1. Age 18 years and older
2. Must sign an informed consent approved by the UAMS Institutional Review Board (IRB)
3. Lung cancer with planned resection.

Cohort E (lung cancer with planned resection) Exclusion criteria:

1. Any other significant medical or psychiatric conditions which, in the opinion of the enrolling investigator, may interfere with consent or compliance of the protocol
2. Existing diagnosis or evidence of Hepatits C, Rheumatoid Arthritis or any previous solid organ transplant.

Cohort F (Any solid tumor cancer with radiation therapy) Inclusion criteria:

1. Age 18 years and older
2. Must sign an informed consent approved by the UAMS Institutional Review Board (IRB)
3. Any solid tumor cancer and will receive radiation therapy.

Cohort F (Any solid tumor cancer with radiation therapy) Exclusion criteria:

1. Any other significant medical or psychiatric conditions which, in the opinion of the enrolling investigator, may interfere with consent or compliance of the protocol 3. Existing diagnosis or evidence of Hepatits C, Rheumatoid Arthritis or any previous solid organ transplant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of genomic profile | 15 months
  Genomic changes causing lung cancer evolve over the course of illness. The genetic changes may serve as a biomarker for diagnosis and response to treatment. These changes will be measured in human specimens and co-cultured in mice.

CONTACTS AND LOCATIONS:
Overall Officials: Donald J Johann, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No